CLINICAL TRIAL: NCT03507699
Title: Combination Treatment of Nivolumab, Ipilimumab, Intratumoral CMP-001 and Radiosurgery for Liver Metastases in Colorectal Carcinoma
Brief Title: Combined Immunotherapy and Radiosurgery for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Checkmate Pharmaceuticals (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Dr. Yaacov Lawrence, Vice Chair, and Director, Center for Translational Research in Radiation Oncology Dep. Radiation Oncology, Sheba Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4465-17-SMC; CA209-991 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2018-04-09; First posted 2018-04-25 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Neoplasms Malignant; Liver Metastases
Keywords: radiotherapy; radiosurgery; immunotherapy; PD-1; CTLA-4; TLR9
MeSH Terms: conditions — Colonic Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: a phase I inter-patient dose-escalation study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immunotherapy alone (Experimental): Nivolumab will be administered at a dose of 3mg/kg every 2 weeks. Ipilimumab will be administered at a dose of 1mg/kg every 6 weeks. CMP-001 will be administered both into the liver metastasis (once), and also injected subcutaneously (four times, over six weeks) at a dose of 5-10 mg.
  Interventions: Drug: Nivolumab Injection [Opdivo]; Drug: Ipilimumab Injection [Yervoy]; Drug: CMP-001
- Combined radiotherapy and immunotherapy (Experimental): Liver radiation therapy: three treatments to one liver metastasis, administered on alternate days.
  Nivolumab will be administered at a dose of 3mg/kg every 2 weeks. Ipilimumab will be administered at a dose of 1mg/kg every 6 weeks. CMP-001 will be administered both into the liver metastasis (once), and also injected subcutaneously (four times, over six weeks) at a dose of 5-10 mg.
  Interventions: Radiation: Liver radiation therapy; Drug: Nivolumab Injection [Opdivo]; Drug: Ipilimumab Injection [Yervoy]; Drug: CMP-001

INTERVENTIONS:
Radiation: Liver radiation therapy — 21 Gy in three fractions to one liver metastasis
  Other Names: Liver radiosurgery
  Arms: Combined radiotherapy and immunotherapy
Drug: Nivolumab Injection [Opdivo] — administered IV at a dose of 3mg/kg every 2 weeks
Drug: Ipilimumab Injection [Yervoy] — administered IV at a dose of 1mg/kg every 6 weeks
Drug: CMP-001 — A TLR9 agonist, will be administered both into the liver metastasis (three times), and also injected subcutaneously at a dose of 5-10 mg every two weeks.

SUMMARY:
A single institution study to evaluate the safety and tolerability of the combination treatment of nivolumab, ipilimumab, CMP-001 and radiosurgery in patients with metastatic colorectal cancer with liver metastases.

DETAILED DESCRIPTION:
Patients will be treated with radiosurgery to liver metastases (completed by day 1), followed by a priming dose of subcutaneous CMP-001 (day 1 ± 4 days), intratumoral injections of CMP-001 on days 13, 36 and 55, combined with nivolumab 3mg/kg every 2 weeks (start day 15) and ipilimumab 1 mg/kg every 6 weeks (start day 15). From day 71 biweekly subcutaneous injections of CMP-001 will commence. Nivolumab, ipilimumab and subcutaneous injections of CMP-001 will be continued until disease progression or up to 24 months in the absence of disease progression or unacceptable toxicity. Two research biopsies will be taken from a liver metastasis. The first biopsy will be taken during the screening period (pretreatment) and the second one 5 weeks post-radiosurgery (which is 3 weeks post-initiation of nivolumab / ipilimumab). As a safety run-in, the initial cohort of 3-6 patients will not receive radiosurgery. The next cohort will not commence until the last patient from the initial cohort has been followed up for at least 8 weeks post first intratumoral injection. Efficacy endpoints will be based upon a non-irradiated lesion.

ELIGIBILITY:
Inclusion Criteria:

Disease factors

* Histologically- or cytologically-confirmed diagnosis of colorectal cancer (CRC).
* Metastatic or recurrent CRC, deemed surgically or medically unresectable.
* Subjects have received two or more standard available therapies known to prolong survival and for which they would be considered eligible, whether in adjuvant or metastatic setting. Such therapies should include regimens containing oxaliplatin and irinotecan in combination with a fluoropyrimidine, if appropriate (e.g., FOLFOX and FOLFIRI, or their variants). Subjects that are unable to receive oxaliplatin and/or irinotecan due to allergy or hypersensitivity, or due to concerns regarding the side effects of oxaliplatin and/or irinotecan, will be allowed to receive less than two lines of standard therapies prior to enrollment to this study.
* Patients must have at least two liver metastases, separated by ≥2 cm, and measured in at least one dimension (longest diameter) as ≥2 cm by CT/MRI. One of the metastases must be amenable to biopsy and SBRT.

General considerations

* Age ≥18 years.
* ECOG performance status ≤1 (Karnofsky ≥70%, see Appendix A).
* Life expectancy of ≥ 3 months
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count ≥1,500/mcL
* platelets ≥100,000/mcL
* hemoglobin ≥ 9.0 g/dL
* total bilirubin ≤ 1.5 x ULN except subjects with Gilbert Syndrome who must have a total bilirubin level < 3.0 mg/dL).
* AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
* creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 50 mL/min (using the Cockcroft Gault formula)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of treatment.
* Signed Written Informed Consent
* Subjects must have signed and dated an IRB approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.

Exclusion Criteria:

Disease factors / Tumor characteristics

* Has an MSI-H phenotype or a known MMR deficiency.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.

Previous treatments and trials

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 3 weeks of the first dose of treatment.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.° Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

Comorbidities, medications and immune modulation agents

* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with type I diabetes mellitus, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Subjects that require intermittent use of bronchodilators or local steroids, e.g., inhaled or topical steroids, at a dose of less than the equivalent of 10mg prednisone daily, would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results.
* History of allergy or hypersensitivity to any study drug components, to compounds of similar chemical or biologic composition
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Previous stem cell transplant.
* Significant bleeding event within the last 12 months that places the patient at risk for intrahepatic IT injection procedure based on Investigator assessment.
* Anticoagulant or anti-platelet medication that cannot be interrupted prior to CMP-001 intratumoral injection, including:

  * Aspirin that cannot be discontinued for 7 days prior to CMP-001 intratumoral injection.
  * Coumadin that cannot be discontinued for 7 days prior to CMP-001 intratumoral injection.
  * Low molecular weight heparin (LMWH) that cannot be discontinued >24 hours prior to CMP-001 intratumoral injection.
  * Unfractionated heparin (UFH) that cannot be discontinued >4 hours prior to CMP-001 intratumoral injection.
  * Oral direct thrombin inhibitor (dabigatran) or direct Factor Xa inhibitor (rivaroxaban, apixiban, and endoxaban) that cannot be discontinued for 4 days prior to CMP-001 intratumoral injection.
  * NOTE: LMWH or UFH may be used to transition patients on and off of the above anti-coagulants (if deemed appropriate by the treating physician) prior to CMP-001 intratumoral injection as long as the last dose of LMWH is administered >24 hours prior to treatments and last dose of UFH is administered >4 hours prior to treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious dose-limiting treatment-related adverse events as assessed by CTCAE v5.0 | The dose-limiting toxicity period lasts from day 1 until day 42 inclusive
  Dose-Limiting Toxicities (DLTs) are defined below and only include AEs that are considered possibly, probably, or definitely related to the CMP-001, nivolumab or ipilimumab treatments which occur during the first 42 days of therapy, starting from completion of SBRT (day 1).
  The following AEs will be considered DLTs if deemed related to study therapy:
  Hematologic
  * Grade 4 neutropenia
  * Febrile neutropenia, defined as absolute neutrophil count (ANC) <1000/mm3 with a temperature of 38.3 degrees Celsius.
  * Grade 3 neutropenic infection
  * Grade 3 thrombocytopenia with bleeding
  * Grade 4 thrombocytopenia
  Non-hematologic:
  * Grade 3 toxicities (non-laboratory)
  * Grade 3 nausea, vomiting or diarrhea despite maximal medical intervention
  * Grade 4 aspartate aminotransferase (AST) and alanine aminotransferase (ALT) Other (non AST/ALT) non-hematologic G 3 laboratory value if the abnormality leads to overnight hospitalization

SECONDARY OUTCOMES:
Response rate as assessed by RECIST v1.1 | assessed at week 10, week 18, and week 24
  To evaluate the objective tumor response rate (ORR; including complete response, CR, or partial response, PR) from a combination treatment with nivolumab, ipilimumab, CMP-001 and radiosurgery as assessed by RECIST v1.1. Of note, the irradiated and injected lesion will not be used for RECIST v1.1 analysis.
Progression free survival | from time of first dose for 24 months
  To evaluate the progression free survival (PFS) for treatment with a combination of nivolumab, ipilimumab, CMP-001 and radiosurgery defined as the time from first dose until disease progression or death (or date of last documentation of being alive), respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No